CLINICAL TRIAL: NCT00694967
Title: Histologic Evaluation of the Cervix at Risk for Preterm Birth Trial:Medical Versus Surgical Therapy
Brief Title: A Randomized Trial of Cerclage Versus 17 α-Hydroxyprogesterone Caproate for Treatment of a Short Cervix
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis showed no difference in outcome between treatment groups.
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Orion Rust M.D., Lehigh Valley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2003103
Record Dates: First submitted 2008-06-07; First posted 2008-06-11 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Mid Trimester Cervical Shortening
Keywords: short cervix, cervical funneling, spontaneous preterm birth, cerclage, progesterone
MeSH Terms: interventions — 17 alpha-Hydroxyprogesterone Caproate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): McDonald cerclage
  Interventions: Procedure: McDonald cerclage placement
- 2 (Active Comparator): 17 hydroxyprogesterone caproate
  Interventions: Drug: 17 hydroxyprogesterone caproate

INTERVENTIONS:
Procedure: McDonald cerclage placement — Transcervical McDonald cerclage placement
  Arms: 1
Drug: 17 hydroxyprogesterone caproate — Weekly 250mg intramuscular injections
  Arms: 2

SUMMARY:
We hypothesized that weekly intramuscular injections of 17 hydroxyprogesterone caproate(17P) will reduce the number spontaneous preterm births prior to 35 weeks gestation when compared to cerclage therapy. The purpose of this study was to compare medical therapy with 17P to surgical therapy with transvaginal cerclage in patients with an ultrasound diagnosed short cervix and funnel in the mid-trimester.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasonographic evidence of premature dilatation of the internal os
* Prolapse of the chorio-amniotic membranes into the endocervical canal
* Functional cervical length less than 25mm
* Exacerbation of these ultrasound findings with transfundal and/or suprapubic pressure

Exclusion Criteria:

* Any fetal chromosomal or structural anomaly
* Multiple gestation
* Known allergy to progesterone
* Ruptured membranes
* Vaginal bleeding
* Intra-amniotic infection (diagnosed clinically or by amniocentesis)
* Prolapse of endocervical membranes beyond the external cervical os
* Persistent uterine activity accompanied by cervical change
* Obstetrically indicated delivery.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2003-11; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome was spontaneous preterm birth prior to 35 weeks gestation | 11/2003 - 12/2006

SECONDARY OUTCOMES:
Obstetrical complications | 11/2003 - 12/2006
Neonatal morbidity & mortality | 11/2003 --12/2006

CONTACTS AND LOCATIONS:
Overall Officials: Orion Rust, M.D, Principal Investigator — Lehigh Valley Hospital
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States